CLINICAL TRIAL: NCT06483880
Title: The Role of Adjuvant Albendazole After Pulmonary Hydatid Cyst Resection: a Randomised Controlled Trial
Brief Title: The Role of Adjuvant Albendazole After Pulmonary Hydatid Cyst Resection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FMASU MS187/2024
Record Dates: First submitted 2024-06-23; First posted 2024-07-03 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2024-02

CONDITIONS: Pulmonary Hydatid Cyst
MeSH Terms: conditions — Echinococcosis, Pulmonary | interventions — Albendazole

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Albendazole arm (Active Comparator): The administration of albendazole therapy is recommended at a dosage of 15 mg/kg/day, given in two equally split doses per day. This is within two 15-day cycles following surgery.
  Interventions: Drug: Albendazole
- Placebo arm (Placebo Comparator): Patients will receive the placebo, which will be in two equally split doses per day. This is within two 15-day cycles following surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Albendazole — Patients will receive albendazole therapy at the recommended dosage.
  Arms: Albendazole arm
Drug: Placebo — Patients will receive the placebo, which will be starch tablets in the same dosage of albendazole.
  Arms: Placebo arm

SUMMARY:
The aim of this study is to study the role of adjuvant Albendazole after pulmonary hydatid cyst resection versus placebo in reducing recurrence with a short- term follow-up of six months.

DETAILED DESCRIPTION:
Hydatid disease, also referred to as cystic echinococcosis, is a major zoonotic disease with global distribution caused by the larval stage of the Echinococcus parasite, which belongs to the Taeniidae family and Echinococcus genus.

Cystic Echinococcosis is prevalent in several regions across the globe, including Mediterranean countries, southern America, Australia, eastern and northern Africa, as well as the Tibetan terrain of Asia.

Dogs and other members of the canid family serve as definitive hosts, as they harbor adult tapeworms within their intestinal tract and excrete parasite eggs in their feces. The intermediate hosts, which encompass a wide range of mammalian species including humans, can get accidentally infected through the ingestion of eggs via food or water that has been contaminated. Upon ingestion of tapeworm eggs found in the feces of dogs, the embryos are liberated from the eggs, traverse the intestinal mucosa, and disseminate to various organs via the bloodstream. The liver accounting for 60% to 70% of infections, and the lungs, comprising around 20% to 30% of infected cases, are the organs most frequently affected by infection.

Surgery is the gold standard treatment to get rid of a pulmonary hydatid cyst, though in some rare cases chemotherapy may be necessary. Despite claims that very small cysts can disappear on their own, surgery remains the gold standard for treating hydatid cysts. Re-surgery after recurrence is associated with increased operative morbidity and mortality. Surgical intervention may sometimes be required due to the development of complications in patients who receive only medical treatment.

Mebendazole was initially used for the therapeutic treatment of the hydatid cyst. Nevertheless, the drug's uptake from the gastrointestinal tract was poor, prompting its substitution with albendazole, which has better absorption. The drug's activity is enhanced by its metabolite, albendazole sulfoxide, which readily diffuses through the cyst membrane and accumulates in the cyst fluid. It has been shown that adjuvant albendazole treatment is effective in reducing recurrence postoperatively in liver hydatidosis.

The standard care in Ain Shams University Hospitals regarding prescription of albendazole after surgery is surgeon's preference. To the best of our knowledge, there was a gap of knowledge regarding the role of adjuvant Albendazole after pulmonary hydatid cyst resection. So, we will conduct this study.

ELIGIBILITY:
Inclusion Criteria:

1. All patients regardless of age with pulmonary hydatid disease requiring surgical resection.
2. Patients achieving complete resection of pulmonary hydatid disease.
3. Patients with no extra pulmonary hydatid disease.
4. Patients who have received preoperative albendazole.

Exclusion Criteria:

1. Patients with extra pulmonary hydatid disease requiring treatment after pulmonary resection.
2. Patients with incomplete resection of pulmonary hydatid disease.
3. Patients with pulmonary hydatid disease not amenable for resection.
4. Patients with hypersensitivity to Albendazole.
5. Patients with liver dysfunction.
6. Patients refusing to be enrolled in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence of pulmonary hydatid disease | six months
  Recurrence of pulmonary hydatid disease in six months in both groups, assessed by:
  1. Chest X-ray radiography after the 2 weeks.
  2. CT chest in six months and after one year or symptoms requiring CT chest at any timing.

SECONDARY OUTCOMES:
Liver function tests (AST and ALT) between both groups. | Six months
  AST and ALT will be measured in U/L before operation and after completing the two 15-day cycles of Albendazole or Placebo in either group. And after six months in both groups.
Length of hospital stay between both groups. | Six months
In hospital mortality between both groups. | Six months
Financial cost between both groups. | Six months

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospitals, Cairo, Al Abbasiya, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arif SH, Shams-Ul-Bari, Wani NA, Zargar SA, Wani MA, Tabassum R, Hussain Z, Baba AA, Lone RA. Albendazole as an adjuvant to the standard surgical management of hydatid cyst liver. Int J Surg. 2008 Dec;6(6):448-51. doi: 10.1016/j.ijsu.2008.08.003. Epub 2008 Aug 16. PMID 18819855
- [Background] Aydin Y, Ulas AB, Ince I, Kalin A, Can FK, Gundogdu B, Kasali K, Kerget B, Ogul Y, Eroglu A. Evaluation of albendazole efficiency and complications in patients with pulmonary hydatid cyst. Interact Cardiovasc Thorac Surg. 2022 Jan 18;34(2):245-249. doi: 10.1093/icvts/ivab259. PMID 34587626
- [Background] Dehkordi AB, Sanei B, Yousefi M, Sharafi SM, Safarnezhad F, Jafari R, Darani HY. Albendazole and Treatment of Hydatid Cyst: Review of the Literature. Infect Disord Drug Targets. 2019;19(2):101-104. doi: 10.2174/1871526518666180629134511. PMID 29956639
- [Background] Fattahi Masoom SH, Lari SM, Fattahi AS, Ahmadnia N, Rajabi M, NaderiKalat M. Albendazole therapy in human lung and liver hydatid cysts: A 13-year experience. Clin Respir J. 2018 Mar;12(3):1076-1083. doi: 10.1111/crj.12630. Epub 2017 Apr 20. PMID 28319358
- [Background] Rawat S, Kumar R, Raja J, Singh RS, Thingnam SKS. Pulmonary hydatid cyst: Review of literature. J Family Med Prim Care. 2019 Sep 30;8(9):2774-2778. doi: 10.4103/jfmpc.jfmpc_624_19. eCollection 2019 Sep. PMID 31681642
- [Background] Sarkar M, Pathania R, Jhobta A, Thakur BR, Chopra R. Cystic pulmonary hydatidosis. Lung India. 2016 Mar-Apr;33(2):179-91. doi: 10.4103/0970-2113.177449. PMID 27051107
- [Background] Teggi A, Lastilla MG, De Rosa F. Therapy of human hydatid disease with mebendazole and albendazole. Antimicrob Agents Chemother. 1993 Aug;37(8):1679-84. doi: 10.1128/AAC.37.8.1679. PMID 8215283